CLINICAL TRIAL: NCT03303664
Title: Inpatient Multimodal Path to RecOVEry
Acronym: IMPROVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: System-wide implementation of intervention prevented randomized trial design
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00022455
Record Dates: First submitted 2017-08-16; First posted 2017-10-06 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2018-02

CONDITIONS: Pain; Opioid Use
Keywords: opioid; inpatient; pain; multimodal
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPROVE Protocol (Experimental): The intervention is composed of 4 parts: 1) a multidisciplinary team that recommends, develops, approves, monitors the components of the intervention and training? 2) monitoring of medication sedation risk using established scale 3) restriction of medication dispensing via enhanced technology 4) health professional training on multimodality pain management including complementary and alternative therapies.
  Interventions: Other: IMPROVE Protocol
- Usual Care (No Intervention): Treatment of patients in the usual manner based on their diagnosis and resources available at that site.

INTERVENTIONS:
Other: IMPROVE Protocol — Comprehensive pain management protocol
  Arms: IMPROVE Protocol

SUMMARY:
The goal of the proposed study is to develop and implement a comprehensive strategy to address pain management in the inpatient setting while appropriately managing pain and optimizing patient safety in the inpatient setting. This strategy involves developing a new health Information Technology tool in the Omnicell and electronic medical record, implementing a "menu" of pain management and relaxation strategies, and developing educational materials for staff and patients to change the culture of pain management.

DETAILED DESCRIPTION:
The goal of the proposed study is to develop and implement a comprehensive strategy to address pain management in the inpatient setting while appropriately managing pain and optimizing patient safety in the inpatient setting. This strategy involves developing a new health Information Technology tool in the Omnicell and electronic medical record, implementing a "menu" of pain management and relaxation strategies, and developing educational materials for staff and patients to change the culture of pain management.

This intervention will be implemented throughout CHS hospitals, using a stepped wedge design to guide rollout. The initial pilot will be conducted in the trauma inpatient units at Carolinas Medical Center. All patients admitted to the two primary trauma units (11A and 11 Tower) during the pilot study period will be included in the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated in facility as inpatient during the study period will be included in the analysis.

Exclusion Criteria:

* Patients not admitted to facility during the study period will be excluded from the analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
Use of Opioid Overdose Reversal Treatment | Patient's entire length of stay in the hospital, up to 3 months
  Incidence of administration of opioid reversal agent

SECONDARY OUTCOMES:
Pain | Patient's entire length of stay in the hospital, up to 3 months
  Average daily pain scores (VAS)
Oversedation without naloxone | Patient's entire length of stay in the hospital, up to 3 months
  Incidence of patient oversedation (Pasero > 2 or associated diagnosis code)
Multimodal Therapy | Patient's entire length of stay in the hospital, up to 3 months
  Percentage of patients receiving multimodal pain management
Average Daily MME | Patient's entire length of stay in the hospital, up to 3 months
  Morphine Milligram Equivalent Dosing for Opioid Medications

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Hsu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (12):
- United States (12):
  - Carolinas Healthcare System - Stanly, Albemarle, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Carolinas Healthcare System - Mercy, Charlotte, North Carolina
  - Carolinas Healthcare System - Pineville, Charlotte, North Carolina
  - Carolinas Healthcare System - University, Charlotte, North Carolina
  - Carolinas Healthcare System - NorthEast, Concord, North Carolina
  - Carolinas Healthcare System - Kings Mountain, Kings Mountain, North Carolina
  - Carolinas Healthcare System - Lincoln, Lincolnton, North Carolina
  - Carolinas Healthcare System - Union, Monroe, North Carolina
  - Carolinas Healthcare System - Blue Ridge, Morganton, North Carolina
  - Carolinas Healthcare System - Cleveland, Shelby, North Carolina
  - Carolinas Healthcare System - Anson, Wadesboro, North Carolina

IPD SHARING:
Plan to Share IPD: No
No IPD will be made available to other researchers.